CLINICAL TRIAL: NCT06025331
Title: From Cuff Arthropathy to Reverse Shoulder Arthroplasty - a Multicentre Randomized Control Trial (Study 1: Does BIO-RSA Provides Superior Clinical Outcome Compared to Conventional RSA?).
Brief Title: Does BIO-RSA Provides Superior Clinical Outcome Compared to Conventional RSA?
Acronym: CARS-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: Haukeland University Hospital (Other); Sykehuset Telemark (Other Government); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARS-1
Record Dates: First submitted 2023-06-28; First posted 2023-09-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Arthroplasty, Replacement, Shoulder; Shoulder Osteoarthritis
Keywords: Reverse Shoulder Arthroplasty; BIO-RSA; Orthopedic surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and health personnel examining the participants will be blinded. It will not be possible to blind the surgeons due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIO-RSA (Experimental)
  Interventions: Procedure: BIO-RSA
- RSA (Active Comparator)
  Interventions: Procedure: RSA

INTERVENTIONS:
Procedure: BIO-RSA — Bony increased offset-reversed shoulder arthroplasty(BIO-RSA) will be performed.
  Other Names: Bony increased offset-reversed shoulder arthroplasty
  Arms: BIO-RSA
Procedure: RSA — Conventional reversed shoulder arthroplasty(RSA) will be performed.
  Other Names: Reverse shoulder arthroplasty
  Arms: RSA

SUMMARY:
The goal of this clinical trial is to compare two different types of reverse shoulder replacements. Researchers will compare a conventional reverse shoulder replacement with a lateralized reverse shoulder replacement to see if there is a difference in how well the patients function after two years.

DETAILED DESCRIPTION:
Many studies have showed pain relief and improvement in shoulder function following reverse shoulder arthroplasty (RSA), but medialization of the centre of rotation (COR) in RSA may cause complications like limited range of motion (ROM), luxation of the prosthesis, and scapular notching, where the lower part of the scapular neck becomes eroded due to impingement against the humeral component. Joint centre lateralization with a bone transplant placed underneath the glenoid component (BIO-RSA) was introduced to maximize ROM in the prosthetic joint, increase stability and to prevent scapular notching. In recent years it has been claimed that lateralization of the COR with BIO-RSA decreases the risk of the aforementioned complication, but no consensus on when or how to lateralize the COR exists as of today. This knowledge will also be of critical importance when it comes to decision making on how these patients are best treated. Results from this research project is expected to have a significant impact on how these patients are treated in the future, both nationally and internationally.

The purpose of this study is to compare functional results between patients with bony increased offset-reversed shoulder arthroplasty (BIO-RSA) and conventional reverse shoulder arthroplasty (RSA) to investigate if lateralization of the glenosphere yields superior outcomes and fewer complications after 2 years.

This multicenter study will include 130 patients in 4 hospitals scheduled for RSA. Patients will be asked to participate in a blinded RCT, where they are randomly assigned to either BIO-RSA or conventional RSA. Functional results will be measured primarily by the patient-reported outcome measure Western Ontario Osteoarthritis Shoulder (WOOS), but they will also be examined by a physiotherapist and CT imagery will be assessed by a radiologist.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for primary RSA due to OA, massive RC tear, failed RC repair or post-instability osteoarthritis
* Able to read or write Norwegian

Exclusion Criteria:

* Severe osteoporosis
* Osteonecrosis of the humeral head
* Dementia
* Poor deltoid function
* Revision surgery
* ASA IV
* Suspected chronic infection
* Acute fracture

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2033-08-01 (Estimated); Study Completion 2033-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in WOOS index from baseline to 24 months postoperatively. | Before randomization, 24 months postoperatively. Also measured 3 and 12 months postoperatively. Change after 24 months will be the primary outcome.
  The Western Ontario Osteoarthritis of the Shoulder (WOOS) index is a patient-reported, disease-specific questionnaire for the measurement of the quality-of-life in patients with osteoarthritis.
  There are 19 questions divided into four domains: Physical symptoms, sports and work, lifestyle and emotions. Each question is answered on a visual analogue scale ranging from 0 to 100. The overall score ranges from 0 to 1900, with 1900 being the worst. For ease of interpretation, the scores are often converted to a percentage of the maximum score.

SECONDARY OUTCOMES:
Change in EuroQol-5 from baseline to 24 months postoperatively. | Before randomization, 3, 12 and 24 months postoperatively.
  The widely used EuroQol-5 (EQ-5D-5L) will be used to measure health-related quality of life.
  The EQ5D-5L consists of two parts: A descriptive system (Mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and the EQ-VAS that record patients self-rated health on a visual analog scale that range from 0 -100, higher levels indicate better self-rated health.
  The descriptive system can be converted to a single summary index number where lower levels indicate poorer health related quality of life.
CT scan | Before randomization, 3, 12 and 24 months postoperatively.
  Assessment of bone transplant integration and fixation of the glenoid implant.
Change in Constant-Murley Score from baseline to 24 months postoperatively. | Before randomization, 3, 12 and 24 months postoperatively.
  The Constant-Murley Score (CMS) is a multi-item functional scale assessing pain, ADL, ROM and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively.
  The test is divided into subjective and objective components. Two subjective: pain and activities of daily living (ADL) and two objective: range of motion (ROM) and strength. The subjective components can receive up to 35 points and the objective 65.
  Pain and ADL are answered by the patient; ROM and strength require a physical evaluation and are answered by the physiotherapist.
Change in range of motion from baseline to 24 months postoperatively. | Before randomization, 3, 12 and 24 months postoperatively.
  The patient's active and passive range of motion (ROM) in the affected shoulder will be measured by an experienced physiotherapist with a long-legged goniometer. The directions measured will be flexion, abduction, external rotation and internal rotation, measured in degrees and/or physical landmarks.
Change in Subjective Shoulder Value from baseline to 24 months postoperatively. | Before randomization, 3, 12 and 24 months postoperatively.
  The Subjective Shoulder Value (SSV) score is defined as the subjective evaluation by the patient of shoulder function, expressed as a percentage of an entirely normal shoulder, which would score 100%.
Anchor question 1 | Before randomization, 3, 12 and 24 months postoperatively.
  This anchor question is asked to help determine Patient Acceptable Symptom State (PASS).
  PASS "Considering all daily activities that involves your operated shoulder, your level of pain and degree of function, how satisfied are you with the condition of your shoulder is right now?" Alternatives: Satisfied/somewhat satisfied/Neither satisfied or unsatisfied/somewhat unsatisfied/Unsatisfied
Anchor question 2 | 3, 12 and 24 months postoperatively.
  This anchor question is asked to help determine Minimal Important Difference (MID) and Substantial Clinical Benefit (SCB).
  "Think of all the ways your operated shoulder has affected you the last week. Since your surgery, has there been any change in the condition of your shoulder that you would consider important or meaningful to you?" Alternatives: Much better/moderately better/a bit better/no change/a bit worse/moderately worse/Much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Sigbjørn Dimmen, PhD, Principal Investigator — University of Oslo; Kjersti Kaul Jenssen, PhD, Principal Investigator — Lovisenberg Diaconal Hospital; Christian Owesen, PhD, Study Director — Lovisenberg Diaconal Hospital
Locations (2):
- Norway (2):
  - Sykehuset Telemark HF, Skien, Telemark
  - Lovisenberg Diaconal Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No